CLINICAL TRIAL: NCT07348211
Title: An Open-Label, Multicenter, First-in-Human Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of SIM0610 in Adult Subjects With Locally Advanced/Metastatic Solid Tumors
Brief Title: First in Human Study of SIM0610 in Solid Tumors
Acronym: SIM0610-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianwei Medical Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0610-101
Record Dates: First submitted 2025-12-24; First posted 2026-01-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumours; Non-Small Cell Lung Cancer; Colorectal Cancer; Head and Neck Squamous Cell Carcinoma; Hepatocellular Carcinoma
Keywords: Locally Advanced/Metastatic Solid Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): SIM0610 administered intravenously at selected dose levels according to protocol
  Interventions: Drug: SIM0610 for Injection
- Cohort expansion (Experimental): SIM0610 administered intravenously at Recommended dosage(RDs) according to protocol
  Interventions: Drug: SIM0610 for Injection

INTERVENTIONS:
Drug: SIM0610 for Injection — intravenous infusion
  Arms: Cohort expansion
Drug: SIM0610 for Injection — intravenous infusion
  Arms: Dose escalation

SUMMARY:
This is a multicenter, open-label, first-in-human (FIH) study to evaluate the safety, tolerability, pharmacokinetic/pharmacodynamic profile, and preliminary antitumor activity of SIM0610 in subjects with locally advanced/metastatic solid tumors. Accelerated titration (ATD) and Bayesian optimal interval design (BOIN) will be used to guide dose escalation in part1, the preliminary anti-tumor effect of SIM0610 will to be further evaluated in part 2.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate and sign the informed consent form
* At least 18 years old, male or female
* Subjects with locally advanced/metastatic solid tumors confirmed by histology and/or cytology;
* Subjects in Part 1 should have at least one tumor lesion evaluable by RECIST v1.1 criteria, and subjects in Part 2 should have at least one measurable tumor lesion by RECIST v1.1 (lesions that have received radiotherapy or other local treatments cannot be used as target lesions unless there is clear progression of the lesion)
* Subjects with locally advanced/metastatic solid tumors who have failed standard treatment: Part 1: Subjects with solid tumors who have experienced disease progression during/after at least one previous standard systemic anti-tumor regimen and are not suitable for standard treatment. Part 2: Non-small cell lung cancer, liver cancer, head and neck squamous cell carcinoma, colorectal cancer that have experienced disease progression during/after at least one previous standard systemic anti-tumor regimen and are not suitable for standard treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Expected survival period ≥ 12 weeks
* Adequate organ and bone marrow function
* Archived formalin-fixed, paraffin-embedded (FFPE) tumor tissue or fresh biopsy tissue within 5 years must be provided before the first administration

Exclusion Criteria:

* A history of active second primary malignancy within the past 2 years, except for localized tumors that are considered cured and have a low risk of recurrence as assessed by the investigator.
* Symptomatic central nervous system (CNS) metastases occurring within 2 weeks prior to the first dose of study treatment; or requirement for local therapy (e.g., radiotherapy or surgery) for CNS metastases; or requirement for corticosteroid therapy for CNS metastases.
* A history of non-infectious interstitial lung disease (ILD)/pulmonary inflammation requiring corticosteroid treatment; current ILD/pulmonary inflammation; or suspected ILD/pulmonary inflammation that cannot be ruled out by screening imaging.
* Uncontrolled pleural effusion, pericardial effusion, or ascites, or occurrence of such effusions requiring drainage or medical intervention within 4 weeks prior to the first dose of study treatment.
* Failure to recover from adverse events (AEs) induced by prior anti-tumor therapy (i.e., recovery to Grade 1 or baseline level).
* Current participation in a study involving investigational drugs or medical devices, or participation in such a study within 4 weeks prior to the first dose of study treatment.
* Receipt of the following therapies prior to the first dose of study treatment:

  1. Cytotoxic therapy within 3 weeks; or anti-tumor targeted small-molecule drugs (e.g., tyrosine kinase inhibitors) within 2 weeks.
  2. Anti-tumor antibody-based immune checkpoint inhibitors, antibody-drug conjugates (ADCs), or other anti-tumor biologics within the shorter of 5 half-lives or 4 weeks.
  3. Traditional Chinese medicines (TCMs)/herbal preparations with anti-tumor indications within 2 weeks.
  4. Radiotherapy within 4 weeks.
* Received antibody-drug conjugate (ADC) with topoisomerase I inhibitor (TOP1i) or other ADC targeting EGFR/cMET.
* Received any live vaccine within 4 weeks prior to the first dose of study treatment.
* Received the following medications ≤ 14 days prior to the first dose of study treatment:

  1. Strong or moderate CYP3A4 induction/inhibitor;
  2. Drugs known to be at risk for torsade de pointes (TdP);
  3. Drugs associated with QTcF interval prolongation (TdP risk equivocal).
* Known human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS).
* A history of clinically significant cardiovascular diseases within 6 months prior to the first dose of study treatment, including but not limited to myocardial infarction, severe/unstable angina pectoris, primary cardiomyopathy, cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction) or congestive heart failure (New York Heart Association [NYHA] Functional Classification > Class II); symptomatic coronary artery disease requiring pharmacotherapy.
* A history of allogeneic organ transplantation or graft-versus-host disease (GVHD).
* A history of hypersensitivity to the active ingredients, inactive excipients of SIM0610, or drugs with similar chemical structures or classifications to SIM0610.
* Pregnant or lactating women. For women of childbearing potential (WOCBP), they are also excluded unless:

  1. The result of serum pregnancy test within 72 hours prior to the first dose of study treatment is negative;
  2. They use highly effective contraceptive methods from the time of signing the informed consent form (ICF) until 180 days after the last dose of study treatment.
* Male subjects with female partners of childbearing potential are excluded unless they use highly effective contraceptive methods from the time of signing the ICF until 180 days after the last dose of study treatment.
* Any other conditions that may increase subject-related risks or interfere with the interpretation of study results, and that, in the investigator's judgment, render the subject unsuitable for study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | From time of first dose of SIM0610 to end of DLT period (approximately 21 days)
Safety and Tolerability | From time of Informed Consent to 28 days post last dose of SIM0610
Objective response rate (ORR) | From date of first dose of SIM0610 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years)
  Objective response rate (ORR) assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - the First Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Cancer Hospital of Shandong First Medical University& Shan Dong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No